CLINICAL TRIAL: NCT02103699
Title: A Prospective Observational Study to Examine Patient Characteristics, Health Care Management, and Effectiveness Among HCV Patients Treated With Simeprevir at Various Practice Settings
Brief Title: A Study to Examine Patient Characteristics, Health Care Management and Health Outcomes of Hepatitis C Virus (HCV) Patients Treated With Simeprevir
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR101973; TMC435HPC4003 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2014-02-18; First posted 2014-04-04 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C virus; Simeprevir; Ribonucleic acid; Sustained virologic response
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis C virus infected patients receiving simeprevir
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Patients receiving simeprevir (single capsule of 150 mg once daily) as prescribed by the health care provider will be observed.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a simeprevir-containing hepatitis C virus (HCV) treatment regimen as measured by sustained virologic response (SVR).

DETAILED DESCRIPTION:
This is a multicenter, observational (a study in which the investigators/ physicians observe the patients and measure their outcomes), prospective study (a study in which the patients are identified and then followed forward in time for the outcome of the study) designed to reflect routine clinical practice. Approximately 300 Hepatitis C virus (HCV) infected patients who are prescribed simeprevir by their health care provider as part of their routine HCV treatment regimen, inclusive of patients who have been treated with a simeprevir-based therapy for less than or equal to (<=) 28 days will be enrolled in this and observed to evaluate the effectiveness of a simeprevir. Practice setting features will be documented at the initiation of the study by each participating site. The decision of patients to participate in this study will in no way impact upon the standard of care that they are receiving. All treatment decisions will be made at the discretion of the health care provider. Safety assessments will include assessment of adverse events, and clinical laboratory parameters (hematology, clotting tests, human immunodeficiency virus tests, chemistry, and liver function tests). The maximum study duration for each patient will be approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have genotype 1 chronic hepatitis C infection
* Hepatitis C virus (HCV) ribonucleic acid (RNA) test result above the limit of quantification before initiation of simeprevir-based therapy
* Health care provider decision to treat patient with a simeprevir-based therapy, inclusive of patients who have been treated with a simeprevir-based therapy for less than or equal to (<=) 28 days will be enrolled into the study
* Prior HCV treatment must be completed more than 3 months before initiation of simeprevir-based therapy
* In the opinion of the health care provider, the patient will attend routine standard of care visits, either at enrolled site or by virtual/telemedicine

Exclusion Criteria:

* Non-genotype 1 HCV infected patients
* Absolute contraindication to any component of prescribed HCV treatment per prescribing information
* Patient is currently enrolled in an interventional study
* Past use of an HCV direct-acting antiviral therapy
* Any investigational drug use within 30 days before initiation of simeprevir-based therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis C virus (HCV) infected patients receiving simeprevir.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients who Achieve Sustained Virologic Response(SVR) | 12 weeks after the actual end of treatment (an expected average of up to 2 years)
  SVR is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) undetectable at least 12 weeks after the actual end of all HCV treatment. Actual end of treatment will be determined by health care provider.

SECONDARY OUTCOMES:
Determination of Prognostic Factors of Virologic Response | 12 weeks after the actual end of treatment (an expected average of up to 2 years)
  Prognostic factors of virologic response includes patient and disease characteristics, treatment paradigm, Rapid Virologic Response (RVR), and select practice setting features. Actual end of treatment will be determined by health care provider.
Total duration of therapy | Up to actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients who Discontinue Therapy by reason | Up to actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients who Achieve Rapid Virologic Response (RVR) | Week 4
  RVR is defined as undetectable hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 4.
Number of Patients who Achieve Sustained Virologic Response(SVR) Among Participants who Achieve Rapid Virologic Response (RVR) | 12 weeks after the actual end of treatment (an expected average of up to 2 years)
  SVR is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) undetectable at least 12 weeks after the actual end of all HCV treatment. RVR is defined as undetectable HCV RNA at Week 4. Actual end of treatment will be determined by health care provider. Actual end of treatment will be determined by health care provider.
Number of Patients who Achieve Sustained Virologic Response(SVR) According to Patient Demographics, Baseline Disease Characteristics, Treatment Paradigm, and Select Practice Setting Features | 12 weeks after the actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients With On-treatment Virologic Failure | Up to actual end of treatment (an expected average of up to 2 years)
  On-treatment virologic failure is defined as a confirmed increase of >1 log10 IU/mL in hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached, or a confirmed HCV RNA level of >100 IU/mL in patients whose HCV RNA had previously been <25 IU/mL. Actual end of treatment will be determined by health care provider.
Number of Patients With Viral Relapse | Up to actual end of treatment (an expected average of up to 2 years)
  Viral Relapse is defined as detectable hepatitis C virus (HCV) ribonucleic acid (RNA) after concluding treatment with undetectable HCV RNA. Actual end of treatment will be determined by health care provider.
Number of Patients With Adverse Events by Grade and Causality | Up to 24 weeks after the actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients With Changes in Clinical Laboratory Parameters by Grade and Causality | Up to 24 weeks after the actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients With Adverse Event Determined to be Related to Simeprevir | Up to 24 weeks after the actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients With Serious Adverse Event | Up to 24 weeks after the actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.
Number of Patients who Develop Mutations at the Time of Virologic Failure | Up to actual end of treatment (an expected average of up to 2 years)
  Actual end of treatment will be determined by health care provider.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (32):
- United States (32):
  - Phoenix, Arizona
  - Bakersfield, California
  - Beverly Hills, California
  - Los Angeles, California
  - Daytona Beach, Florida
  - DeLand, Florida
  - Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Crestview Hills, Kentucky
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Newark, New Jersey
  - Vineland, New Jersey
  - Brooklyn, New York
  - Flushing, New York
  - New York, New York
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Rocky Mount, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Doylestown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Murray, Utah
  - Norfolk, Virginia